CLINICAL TRIAL: NCT02227121
Title: Acute Defibrillation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient enrollments under current protocol for further development & studies
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASD Study
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Ventricular Arrhythmias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VT/VF induction and defibrillation (Experimental): Ventricular Tachycardia and Ventricular Fibrillation (VT/VF) induction and defibrillation will be carried out as the invention in all subjects undergoing study procedures.
  Interventions: Device: Defibrillation following induction of VT/VF

INTERVENTIONS:
Device: Defibrillation following induction of VT/VF — Up to 10 VT/VF induction attempts followed by shock(s) delivered by an externally placed ICD and/or external defibrillator.

SUMMARY:
The proposed study is designed to characterize defibrillation efficacy in humans for the potential development of a new extravascular implantable cardioverter defibrillator (ICD) system.

DETAILED DESCRIPTION:
The study recruited male and female subjects that met all of the inclusion criteria and none of the exclusion criteria. All subjects were scheduled to undergo surgical procedures outlined in the inclusion criteria. These surgical procedures were chosen as the patient population for this study because these procedures require similar personnel and may require access to similar or the same spaces as the ASD procedure.

The entire ASD study research system was removed prior to proceeding with the subject's planned surgery per standard medical practice, which then proceeded according to the standard of care.

Subjects were followed through their routine post-surgery follow-up visit.

At the time of completing the follow-up visit, the subjects' participation was complete and the subjects exited the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be undergoing surgical procedure for approved indications for
* cardiothoracic surgery where a midline sternotomy is planned, or
* implant of a transvenous (TV) ICD or subcutaneous ICD (S-ICD®), or
* VT ablation procedure, or
* VT inducibility testing during Electrophysiology (EP) study
* Subject must be willing to provide Informed Consent
* Subject must be ≥ 18 years old

Exclusion Criteria:

* Subject is considered to be at high risk for infection
* Subject has Left Ventricular Ejection Fraction (LVEF) ≤ 20%
* Subject at high risk of stroke
* Subject with an implanted active cardiac or non-cardiac device during study procedure (e.g., ICD, S-ICD®, Pacemaker, Neuro stimulator)
* Subject is pacemaker dependent
* Subject had previous pericarditis or prior sternotomy
* Subject has hiatus hernia or moderate or worse pectus excavatum
* Subject has hypertrophic cardiomyopathy
* Subject has severe aortic stenosis
* Subject has severe proximal three vessel coronary disease (over 70% in each vessel)
* Subject has >50% left main stem (LMS) disease
* Subject has known skin irritations to the Physio Control Fast Patch ECG Electrode
* Subject is enrolled in a concurrent study that may confound the results of this study, without documented pre-approval from a Medtronic study manager
* Subject has medical conditions that would limit study participation
* Subject is pregnant
* Subject meets exclusion criteria required by local law (e.g. age, breast feeding, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
- Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow, Poland
- United Kingdom (3):
  - Liverpool Heart and Chest Hospital, Liverpool
  - King's College Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Subjects: All subjects consented for the study.
Period: Overall Study
Arm/Group | Enrolled Subjects
Started (Subject underwent attempted VF induction during surgery procedure) | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 61.6 [54 to 70.5]
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom: Hong Kong | 7
  United Kingdom: United Kingdom | 5
  United Kingdom: Poland | 3
  United Kingdom: Netherlands | 1
Primary Indication for Surgery [Count of Participants; unit: Participants]
  Cardiac Surgery: Coronary Artery Bypass Graft | 2
  Cardiac Surgery: Valve Replacement | 5
  Cardiac Surgery: Valve Repair | 2
  Surgery Related to ICD (transvenous) | 1
  Surgery Related to S-ICD (subcutaneous ICD) | 5
  Aortic Aneurysm | 1

OUTCOME MEASURES:

1. Primary Outcome: Defibrillation Outcome
Description: Subjects will demonstrate a successful defibrillation outcome if they have a successful defibrillation shock with the research system.
Time Frame: Day of procedure
Population: Only subjects with ventricular fibrillation successfully induced were eligible for analysis
Measure: Count of Participants; unit: Participants
Groups:
- VF Induction and Defibrillation: Ventricular Fibrillation (VF) induction and defibrillation will be carried out as the invention in all subjects undergoing study procedures.
  Defibrillation following induction of VF: Up to 10 VF induction attempts followed by shock(s) delivered by an externally placed Implantable Cardioverter/Defibrillator (ICD) and/or external defibrillator.
Arm/Group | VF Induction and Defibrillation
Number analyzed (Participants) | 14
Participants
  VF Successfully Terminated with 35J shock | 13
  VF Not Successfully Terminated with 35J shock | 1
Statistical Analysis 1: Comparison: VF Induction and Defibrillation; Null Hypothesis: Percentage of Subjects with Successful VF Termination ≤ 65% Alternative Hypothesis: Percentage of Subjects with Successful VF Termination > 65%; Test type: Superiority or Other; Percentage = 92.86, 95% CI 1-sided [lower limit 70.3]

ADVERSE EVENTS:
Time Frame: Baseline Assessment to routine Post-surgery follow-up visit.
Groups:
- Enrolled Subjects: All subjects consented into the study
Arm/Group | Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=16)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=16)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Post-traumatic headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.